CLINICAL TRIAL: NCT02833727
Title: Assessment of Airway Inflammation and Disease Burden in Moderate to Severe Asthmatic Smokers
Brief Title: Airway Inflammation and Disease Burden in Asthmatic Smokers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Montréal (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, Catherine Lemiere, MD,MSc, Université de Montréal
Other Study IDs: 2017-1359
Record Dates: First submitted 2016-07-07; First posted 2016-07-14 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Asthma
Keywords: asthma; smoking; Eosinophils; health care costs
MeSH Terms: conditions — Asthma; Smoking | interventions — Smoking Devices

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthmatic smokers (AS): Asthmatics will fulfill the following definition of asthma: reversible airflow obstruction and/or a provocative concentration of methacholine inducing a 20% fall in FEV1 (PC20) < 8 mg/ml with a diagnosis of asthma made by a respirologist.
  Smokers or ex smokers will be defined by a smoking history of ≥ 10 pack/year.
  Interventions: Other: Smoking
- Asthmatic non-smokers (ANS): Asthmatics will fulfill the following definition of asthma: reversible airflow obstruction and/or a PC20 < 8 mg/ml with a diagnosis of asthma made by a respirologist.
  Never smokers will have a life-long history without smoking.
  Interventions: Other: Smoking

INTERVENTIONS:
Other: Smoking — Smoking equal or greater than 10 pack/years; never smokers: lifelong history without smoking.

SUMMARY:
Aim : To compare, among patients with an uncontrolled moderate to severe asthma, the blood eosinophil levels of smokers and non-smokers.

Secondary aims: In uncontrolled moderate to severe asthmatic subjects, to compare between asthmatic smokers and non-smokers: sputum eosinophils counts, fractional exhaled nitric oxide (FeNO), pre and post bronchodilator Forced expiratory volume in one second (FEV1) / Forced vital capacity (FVC), Asthma-related quality of life, asthma exacerbations during the year preceding enrolment in the study, Medical direct and indirect costs related to asthma during the year preceding enrolment in the study, and adherence to asthma treatment during the year preceding enrolment in the study.

Methods: Cross sectional observational study. Never-smoker and smoker asthmatics treated with at least 2 controller medications with a smoking history ≥10 pack/year with a ACQ score ≥ 1.5 points will be identified in the database RESP. Their clinical data will be matched to the Régie de l'assurance médicale du Quebec (RAMQ) and Maintenance et exploitation des données pour l'étude de la clientèle hospitalière (MED-ECHO) administrative databases and reMed (data on medications for patients with private health insurance) in order to access to data on medical services, hospitalisations and medications delivered by pharmacies. T

DETAILED DESCRIPTION:
Aim : To compare, among patients with an uncontrolled moderate to severe asthma, the blood eosinophil levels of smokers and non-smokers.

Hypothesis: Uncontrolled never-smoker asthmatics (NSA) will have a greater level of blood eosinophils than uncontrolled asthmatic smokers (AS) (difference in blood eosinophil count at least superior to 100 eosinophils per μL).

Secondary aims: In uncontrolled moderate to severe asthmatic subjects, to compare between asthmatic smokers and non-smokers: sputum eosinophils counts, fractional exhaled nitric oxide (FeNO), pre and post bronchodilator FEV1 / Forced vital capacity (FVC), Asthma-related quality of life, asthma exacerbations during the year preceding enrolment in the study, Medical direct and indirect costs related to asthma during the year preceding enrolment in the study, and adherence to asthma treatment during the year preceding enrolment in the study.

Methods: Cross sectional observational study. Never-smoker and smoker asthmatics treated with at least 2 controller medications with a smoking history ≥10 pack/year with a ACQ score ≥ 1.5 points will be identified in the Quebec registry in respiratory health (RESP). Their clinical data will be matched to the "Régie de l'assurance médicale du Quebec" (RAMQ) and "Maintenance et exploitation des données pour l'étude de la clientèle hospitalière" (MED-ECHO) administrative databases and database on medications dispensed in community pharmacies to patients with private drug insurance (reMed) in order to access to data on medical services, hospitalisations and medications delivered by pharmacies. The subjects identified in the RESP database fulfilling the definition of moderate to severe uncontrolled asthma will be contacted. The Asthma Control Questionnaire (ACQ) will be administered to the subjects over the phone. Subjects with an ACQ score ≥ 1.5 points will be invited to come to the research center of Sacré-Coeur Hospital. During a unique visit at the Hospital du Sacré-Coeur de Montréal, after signature of the consent form, 80 asthmatic smokers and 80 non-smoker asthmatic subjects will be asked to complete questionnaires regarding asthma control (if the delay between telephone interview and visit to the hospital exceed one week), quality of life, and asthma impact on daily activities. FeNO will be measured first. They will then perform spirometry. Sputum induction will be performed to obtain sputum cell counts. Blood will be drawn to obtain blood eosinophil count and serum cotinine. We will be able to compare between asthmatic smokers and non-smoker asthmatics: blood eosinophil counts, sputum eosinophils counts, FeNO, pre and post bronchodilator FEV1 / FVC, asthma-related quality of life, asthma exacerbations during the year preceding enrolment in the study, Medical direct and indirect costs related to asthma during the year preceding enrolment in the study, and adherence to asthma treatment during the year preceding enrolment in the study.

Significance: Anti-interleukin 5 have been shown to be very effective in reducing asthma exacerbations in asthmatic subjects with eosinophilic inflammation with frequent asthma exacerbations. However, smokers have been excluded from these studies. It will be important to determine the burden of asthma in this group of subjects in term of healthcare utilization and productivity at work, in order to evaluate whether or not they may benefit from this type of medication. If we show that the direct and indirect cost related to asthma are higher in asthmatic smokers than non-smokers, it will be even more important to characterize the airway inflammation of this group of subjects in order to determine whether they are likely candidates to receive new biologic agents in order to improve asthma control, decrease their healthcare utilization and improve their productivity at work.

ELIGIBILITY:
Inclusion Criteria:

* Participation to the RESP Database.
* Never-smoker and smoker asthmatics (smoking history ≥10 pack/year)
* Treatment with at least 2 controller medications
* ACQ score ≥ 1.5 points will be identified in the database RESP.

Exclusion Criteria:

* Chronic obstructive Pulmonary Disease (COPD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Never-smoker and smoker asthmatics treated with at least 2 controller medications with a smoking history ≥10 pack/year with a ACQ score ≥ 1.5 points
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
blood eosinophil count | one year

SECONDARY OUTCOMES:
Sputum eosinophil count | One year
Fractional exhaled nitric oxide (FeNO) | One year
FEV1 | One year
Asthma-related quality of life score | One year
  We will use the Asthma Quality of Life Questionnaire (AQLQ). This is a 32-item, self-administered, disease-specific quality of life questionnaire that evaluates asthma quality of life across 4 domains: activity limitation, symptoms, emotional distress, and environmental stimuli. Each item is rated on a 7-point scale (1=maximal impairment, 7=no impairment) to yield a mean score out of 7.
Asthma exacerbations | Two years
Medical direct and indirect costs related to asthma | Two years
Adherence to asthma treatment measured by the proportion of days covered (PDC)(%) | Two years
  Adherence to controller medications will be measured with the proportion of days covered (PDC), a widely used measure of adherence based on prescription claims data. The PDC will be defined as the sum of the duration of all prescriptions of the medication under study filled in the year preceding the visit, divided by 365 days, expressed in percent. The PDC will be estimated using prescription refills data obtained from the RAMQ and reMed databases in the year preceding enrolment.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lemiere, MD, Principal Investigator — CIUSS du nord de l'île de Montréal
Locations (1):
- Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tan NC, Nguyen HV, Lye WK, Sankari U, Nadkarni NV. Trends and predictors of asthma costs: results from a 10-year longitudinal study. Eur Respir J. 2016 Mar;47(3):801-9. doi: 10.1183/13993003.00188-2015. Epub 2015 Dec 2. PMID 26647437
- [Background] Chaudhuri R, Livingston E, McMahon AD, Thomson L, Borland W, Thomson NC. Cigarette smoking impairs the therapeutic response to oral corticosteroids in chronic asthma. Am J Respir Crit Care Med. 2003 Dec 1;168(11):1308-11. doi: 10.1164/rccm.200304-503OC. Epub 2003 Jul 31. PMID 12893649
- [Background] Sunyer J, Springer G, Jamieson B, Conover C, Detels R, Rinaldo C, Margolick J, Munoz A. Effects of asthma on cell components in peripheral blood among smokers and non-smokers. Clin Exp Allergy. 2003 Nov;33(11):1500-5. doi: 10.1046/j.1365-2222.2003.01730.x. PMID 14616860